CLINICAL TRIAL: NCT02387216
Title: SHERLOC: A Phase 2 Study of MM-121 in Combination With Docetaxel Versus Docetaxel Alone in Patients With Heregulin Positive, Locally Advanced or Metastatic Non-Small Cell Lung Cancer (Merrimack Pharmaceuticals Inc.)
Brief Title: A Study of MM-121 in Combination With Chemotherapy Versus Chemotherapy Alone in Heregulin Positive NSCLC
Acronym: SHERLOC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on the preliminary results seen during interim analysis, which were confirmed in the final analysis, the Sponsor terminated the study
Sponsor: Elevation Oncology (Industry)
Collaborators: Merrimack Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM-121-01-02-09
Record Dates: First submitted 2015-02-12; First posted 2015-03-12 (Estimated); Results first posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Non-Small Cell Lung Cancer; NSCLC; Adenocarcinoma; Heregulin
Keywords: NSCLC; Non-Small Cell Lung Cancer; heregulin; ErbB3; docetaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma; Fibromatosis, Gingival, 2 | interventions — seribantumab; Docetaxel

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, international, multi-center, Phase 2 study in patients with locally advanced or metastatic non-small cell lung cancer (NSCLC)
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Experimental Arm (Experimental): MM-121 in combination with Docetaxel
  Interventions: Drug: MM-121; Drug: Docetaxel
- Arm B: Comparator Arm (Active Comparator): Docetaxel alone
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: MM-121 — Investigational, fully human antibody targeting and inhibiting ErbB3
  Other Names: seribantumab
  Arms: Arm A: Experimental Arm
Drug: Docetaxel — approved chemotherapy treatment for NSCLC
  Other Names: Taxotere

SUMMARY:
The purpose of this study is to determine whether the combination of MM-121 plus docetaxel is more effective than docetaxel alone in regards to PFS in patients with heregulin-positive NSCLC.

DETAILED DESCRIPTION:
This study is a randomized, open-label, international, multi-center, phase 2 study in patients with Heregulin-positive NSCLC histologically classified as adenocarcinoma that have progressed following no more than two systemic therapies for locally advanced or metastatic disease, one of which must have been a platinum containing regimen. All patients will initially be screened for heregulin status. Eligible patients will be randomized to receive MM-121 in combination with docetaxel versus docetaxel alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of cytologically or histologically documented adenocarcinoma of the lung with either metastatic disease (stage IV), Stage IIIB or Stage IIIC disease not amenable to surgery with curative intent
* Not received more than 2 prior systemic therapies- one of which must have been a platinum based regimen- for primary or recurrent disease
* Tissue submitted for HRG-biomarker testing
* ECOG performance status (PS) of 0 or 1

Exclusion Criteria:

* Known ALK mutation
* Presence of exon 19 deletion or exon 21 (L858R) substitution of the EGFR gene
* Received >2 prior systemic anti-cancer drug regimen for locally advanced disease
* Prior treatment with an anti-ErbB3 antibody
* CTCAE grade 3 or higher peripheral neuropathy
* Symptomatic CNS metastases or CNS metastases requiring steroids
* Any other active malignancy requiring systemic therapy
* Clinically significant cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MM-121 Program Medical Director, MD, Study Director — Merrimack Pharmaceuticals
Locations (32):
- United States (15):
  - Tucson, Arizona
  - Los Angeles, California
  - Santa Rosa, California
  - Tampa, Florida
  - Chicago, Illinois
  - Lafayette, Indiana
  - Boston, Massachusetts
  - Danvers, Massachusetts
  - New York, New York
  - The Bronx, New York
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Nashville, Tennessee
  - Fairfax, Virginia
  - Seattle, Washington
- Toronto, Ontario, Canada
- France (2):
  - Centre Léon Bérard, Lyon, Auvergne-Rhône-Alpes
  - CHI Creteil, Créteil, Paris
- Germany (5):
  - München, Bavaria
  - Bad Berka
  - Berlin
  - Frankfurt
  - Oldenburg
- Hungary (3):
  - Budapest
  - Miskolc
  - Tatabánya
- Spain (6):
  - Badalona, Barcelona
  - Majadahonda, Madrid
  - Barcelona
  - Madrid
  - Málaga
  - Zaragoza

REFERENCES:
- [Derived] Sequist LV, Gray JE, Harb WA, Lopez-Chavez A, Doebele RC, Modiano MR, Jackman DM, Baggstrom MQ, Atmaca A, Felip E, Provencio M, Cobo M, Adiwijaya B, Kuesters G, Kamoun WS, Andreas K, Pipas JM, Santillana S, Cho BC, Park K, Shepherd FA. Randomized Phase II Trial of Seribantumab in Combination with Erlotinib in Patients with EGFR Wild-Type Non-Small Cell Lung Cancer. Oncologist. 2019 Aug;24(8):1095-1102. doi: 10.1634/theoncologist.2018-0695. Epub 2019 Apr 11. PMID 30975923

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 87 multi-national sites
Pre-assignment Details: One patient was inappropriately enrolled into the sherloc study hence why 152 and not 153
Groups:
- Arm A (Experimental): MM-121 in Combination With Docetaxel: MM-121 (Seribantumab, a human monoclonal antibody that targets ErbB3, a cell surface receptor that is activated by the ligand heregulin. Heregulin-driven ErbB3 signaling has been implicated as a mechanism of tumor growth and resistance to targeted, cytotoxic and anti-endocrine therapies. When used in the combination setting, seribantumab is designed to block ErbB3 signaling in order to enhance the anti-tumor effect of a combination therapy partner): 3000 mg fixed dose intravenous (IV) on Day 1 of each 21-day cycle
  Docetaxel (approved chemotherapy treatment for non-small cell lung cancer (NSCLC)): 75 mg/m˄2 IV on Day 1 of each 21-day cycle
- Arm B (Comparator): Docetaxel Alone: Docetaxel (approved chemotherapy treatment for NSCLC):
  75 mg/m˄2 IV on Day 1 of each 21-day cycle
Period: Overall Study
Arm/Group | Arm A (Experimental): MM-121 in Combination With Docetaxel | Arm B (Comparator): Docetaxel Alone
Started (One patient was inappropriately enrolled into the Sherloc study hence why 152 participants started and not 153) | 103 | 49
Completed (Safety population: includes patients receiving at least one dose of study medication) | 3 | 2
Not Completed | 100 | 47
Not completed — Progressive disease | 2 | 0
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Physician Decision | 2 | 0
Not completed — Sponsor Decision | 28 | 12
Not completed — Death | 60 | 23
Not completed — Other | 5 | 4
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Population: Patients that have signed informed consent, identified as HRG positive based on centralized tissue analysis,& have successfully completed study entry criteria (Safety Population- patients receiving at least one dose of study medication. All safety analyses were performed on either the Modified Intent-to-Treat (mITT) Population or this population).
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Experimental): MM-121 in Combination With Docetaxel | Arm B (Comparator): Docetaxel Alone | Total
Number analyzed (Participants) | 103 | 49 | 152
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 58 | 31 | 89
  >=65 years | 45 | 18 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (10.07) | 62.8 (7.28) | 62.8 (8.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 19 | 51
  Male | 71 | 30 | 101
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 90 | 41 | 131
  Unknown or Not Reported | 7 | 4 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 2 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 83 | 38 | 121
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  Australia | 9 | 3 | 12
  Canada | 2 | 6 | 8
  France | 11 | 6 | 17
  Germany | 7 | 4 | 11
  Hungary | 1 | 1 | 2
  Poland | 2 | 2 | 4
  South Korea | 0 | 1 | 1
  Spain | 28 | 10 | 38
  Taiwan | 2 | 1 | 3
  Thailand | 3 | 0 | 3
  United States | 38 | 15 | 54
Metastatic burden (TNM Stage at Initial Diagnosis) [Count of Participants; unit: Participants] — Based upon the population treated, the most important baseline measure was CT scans to determine metastatic burden, as the primary endpoint was investigator assessed PFS.
  TNM Staging (Tumor size):
  T1 (T1a,T1b & T1c): <3 cm across. T2 (T2a/T2b): > 3 cm but not larger than 5 cm across. T3: > 5 cm but not larger than 7 cm across. T4: Tumor larger than 7cm across. As a rule, the lower the number, the less the cancer has spread. A higher number, such as stage IV, means cancer has spread more. And within a stage, an earlier letter means a lower stage.
  Participants
    Stage IIA | 5 | 3 | 8
    Stage IIB | 1 | 1 | 2
    Stage IIIA | 7 | 4 | 11
    Stage IIIB | 13 | 8 | 21
    Stage IV | 77 | 33 | 110
Heregulin positive status and staining in archival tissue [Count of Participants; unit: Participants] — Measure Description: Patients had to be ≥ HRG 1 positive in their submitted tumor sample to qualify for the study
  Participants | 103 | 49 | 152

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression Free Survival is defined as the time from randomization to the first documented radiographical progression of disease using RECIST v.1.1, or death from any cause, whichever came first based on investigator assessment.
  Patients that do not experience progression or death at the time of analysis were to be progression censored at the date of last valid tumor assessment. Progression-free survival time distribution and median survival for each treatment group were analyzed using the Kaplan-Meier method. Tumor response was evaluated by the local radiologist according to RECIST version 1.1 to establish disease progression by CT or MRI.
Time Frame: Randomization until progression of disease or death due to any cause within 3 years,11 months (the study terminated prematurely)
Population: The Modified Intent-to-Treat (mITT) Population consisted of all randomized patients who received at least 1 dose of assigned therapy
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Arm A (Experimental): MM-121 in Combination With Docetaxel | Arm B (Comparator): Docetaxel Alone
Number analyzed (Participants) | 71 | 38
months | 3.4 [1.9 to 5.7] | 4.1 [2.7 to 6.3]
Statistical Analysis 1: Comparison: Arm A (Experimental): MM-121 in Combination With Docetaxel vs Arm B (Comparator): Docetaxel Alone; Test type: Superiority; p = 0.2302, Log Rank; Hazard Ratio (HR) = 1.382, 95% CI 2-sided [0.813 to 2.350]

2. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) is defined as the time from the date of randomization to the date of death from any cause
Time Frame: From date of randomization until the date of death from any cause assessed upto 3 years,11 months (the study terminated prematurely)
Population: Modified Intent-to-Treat (ITT) population
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Arm A (Experimental): MM-121 in Combination With Docetaxel | Arm B (Comparator): Docetaxel Alone
Number analyzed (Participants) | 71 | 38
months | 7.7 [3.6 to 10.4] | 8.4 [5.8 to 14.7]
Statistical Analysis 1: Comparison: Arm A (Experimental): MM-121 in Combination With Docetaxel vs Arm B (Comparator): Docetaxel Alone; Test type: Superiority; p = 0.5436, Log Rank; Hazard Ratio (HR) = 1.195, 95% CI 2-sided [0.673 to 2.122]

3. Secondary Outcome: Objective Response Rate
Description: Objective Response Rate (ORR) is defined as the proportion of patients a best overall response characterised as either a Complete Response (CR) or Partial Response (PR), as defined according to RECIST v1.1 guidelines, relative to the total number of evaluable patients.
  Complete Response (CR) is defined as disappearance of all lesions and pathologic lymph nodes.
  Partial Response (PR) is defined as >=30% decrease in the sum of the longest diameter of target lesions
Time Frame: Randomization through end of study up to 3 years, 11 months (the study terminated prematurely)
Population: Modified Intent-to-Treat (ITT) population
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Experimental): MM-121 in Combination With Docetaxel | Arm B (Comparator): Docetaxel Alone
Number analyzed (Participants) | 71 | 38
Participants
  Objective Response | 14 | 2
  Partial Response (PR) | 14 | 2
  Stable Disease (SD) | 39 | 26
  Progressive Disease | 12 | 5
  Not Evaluable | 1 | 1
  No Evaluation | 5 | 4
Statistical Analysis 1: Comparison: Arm A (Experimental): MM-121 in Combination With Docetaxel vs Arm B (Comparator): Docetaxel Alone; Test type: Superiority; p = 0.0455, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 4.3

4. Secondary Outcome: Time to Progression
Description: Time to Progression (TTP) is defined as the time from the date of randomization to the date of objective tumor progression. In the actual analysis, duration of response (DOR) was analysed.
Time Frame: Randomization to date of objective tumor progression up to 3 years, 11 months (the study terminated prematurely)
Population: Modified Intent-to-Treat Population
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Arm A (Experimental): MM-121 in Combination With Docetaxel | Arm B (Comparator): Docetaxel Alone
Number analyzed (Participants) | 71 | 38
months | 3.0 [2.8 to 5.2] | NA [NA to NA] — Due to an insufficient number of participants with event
Statistical Analysis 1: Comparison: Arm A (Experimental): MM-121 in Combination With Docetaxel vs Arm B (Comparator): Docetaxel Alone; Test type: Superiority; p = 0.2726, Log Rank

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events Reported With the Combination of MM-121 With Docetaxel Versus Docetaxel Alone
Description: Treatment-emergent adverse events (TEAEs) are defined as any event that occurred after the first dose of study drug and was not present prior to study drug administration or worsened in severity after study drug administration
Time Frame: TEAEs were collected through the study completion (02 Jan 2019), up to 3 years, 11 months
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Arm A (Experimental): MM-121 in Combination With Docetaxel | Arm B (Comparator): Docetaxel Alone
Number analyzed (Participants) | 103 | 49
participants
  Patients with any TEAE-Related | 99 | 45
  Patients with any TEAE-Serious Adverse event | 40 | 15
  Patients with any NCI-CTCAE Grade 3 or Higher | 76 | 31

6. Secondary Outcome: Pharmacokinetic (PK) Parameters of MM-121 in Combination With Docetaxel and Docetaxel When Given in Combination With MM-121.
Description: Pharmacokinetic (PK) profile of MM-121 when given in combination with docetaxel, and of docetaxel when given in combination with MM-121. The maximum observed concentration (Cmax) were to be presented and calculated using non-compartmental analysis. Serum levels of MM-121 were to be measured at a central lab using an enzyme-linked immunosorbent assay.
Time Frame: The study terminated prematurely after 3 years, 11 months (02 Jan 2019). PK evaluation were to be performed on samples obtained at Week 1 pre-dose and post-dose and at pre-dose at Cycle 2 and beyond to assess pre-treatment through concentrations of MM-121
Population: The PK data were not collected for this abbreviated report. There was no pharmacokinetic data feasible for the analysis, and as such, no related analyses were performed. Hence, data could not be reported in the data table.
Arm/Group | Arm A (Experimental): MM-121 in Combination With Docetaxel | Arm B (Comparator): Docetaxel Alone
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events Reported With the Combination of MM-121 With Docetaxel Versus Docetaxel Alone
Description: as for outcome 5
Time Frame: TEAEs were collected through the study completion (02 Jan 2019), up to 3 years, 11 months
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | Arm A (Experimental): MM-121 in Combination With Docetaxel | Arm B (Comparator): Docetaxel Alone
Number analyzed (Participants) | 103 | 49
percentage of participants
  TEAE-Related | 96.1 | 91.8
  TEAE-Serious Adverse event | 38.8 | 30.6
  NCI-CTCAE Grade 3 or Higher | 73.8 | 63.3

ADVERSE EVENTS:
Time Frame: From Baseline through to premature study completion up to 3 years, 11 months (02 Jan 2019)
Description: The safety population includes patients receiving at least one dose of study medication. All safety analyses were be performed on this population. Safety analyses (adverse events and laboratory analyses) were performed using the safety population. Adverse events were coded using the latest MedDRA dictionary (MedDRA 21.0). Severity of adverse events was graded according to the NCI CTCAE version 4.03.
Arm/Group | Arm A (Experimental): MM-121 in Combination With Docetaxel | Arm B (Comparator): Docetaxel Alone
All-Cause Mortality (participants affected / at risk) | 64/103 | 25/49
Serious Adverse Events (participants affected / at risk) | 40/103 | 15/49
Other Adverse Events (participants affected / at risk) | 103/103 | 47/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Experimental): MM-121 in Combination With Docetaxel (N=103) | Arm B (Comparator): Docetaxel Alone (N=49)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 4
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Cardio pulmonary failure (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 0
Colitis (Gastrointestinal disorders) | 3 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 0
Chest pain (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 8 | 1
Sepsis (Infections and infestations) | 1 | 2
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Listeriosis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Lipase increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Starvation (Metabolism and nutrition disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Experimental): MM-121 in Combination With Docetaxel (N=103) | Arm B (Comparator): Docetaxel Alone (N=49)
Anaemia (Blood and lymphatic system disorders) | 29 | 11
Neutropenia (Blood and lymphatic system disorders) | 29 | 11
Febrile neutropenia (Blood and lymphatic system disorders) | 8 | 6
Leukopenia (Blood and lymphatic system disorders) | 6 | 4
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 4 | 0
Sinus tachycardia (Cardiac disorders) | 3 | 2
Atrial flutter (Cardiac disorders) | 2 | 0
Cardio pulmonary failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Cushingoid (Endocrine disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 7 | 4
Dry eye (Eye disorders) | 3 | 0
Blepharospasm (Eye disorders) | 2 | 0
Eye irritation (Eye disorders) | 2 | 0
Vision blurred (Eye disorders) | 2 | 0
Eye pruritus (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 52 | 11
Nausea (Gastrointestinal disorders) | 30 | 14
Stomatitis (Gastrointestinal disorders) | 19 | 2
Vomiting (Gastrointestinal disorders) | 13 | 4
Constipation (Gastrointestinal disorders) | 7 | 7
Dyspepsia (Gastrointestinal disorders) | 6 | 2
Dry mouth (Gastrointestinal disorders) | 5 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 3
Haemorrhoids (Gastrointestinal disorders) | 3 | 1
Abdominal discomfort (Gastrointestinal disorders) | 3 | 0
Colitis (Gastrointestinal disorders) | 3 | 3
Flatulence (Gastrointestinal disorders) | 3 | 0
Abdominal pain lower (Gastrointestinal disorders) | 2 | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Odynophagia (Gastrointestinal disorders) | 2 | 0
Oesophagitis (Gastrointestinal disorders) | 2 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 1
Oral pain (Gastrointestinal disorders) | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Anal inflammation (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Glossitis (Gastrointestinal disorders) | 1 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1
Rectal tenesmus (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 45 | 16
Asthenia (General disorders) | 28 | 11
Mucosal inflammation (Gastrointestinal disorders) | 15 | 5
Pyrexia (General disorders) | 13 | 9
Pain (General disorders) | 8 | 6
Oedema peripheral (General disorders) | 5 | 3
Chills (General disorders) | 4 | 0
Chest pain (General disorders) | 3 | 1
General physical health deterioration (General disorders) | 3 | 1
Oedema (General disorders) | 2 | 5
Non-cardiac chest pain (General disorders) | 2 | 0
Xerosis (General disorders) | 2 | 0
Ulcer (General disorders) | 1 | 1
Cyst (General disorders) | 1 | 0
Extravasation (General disorders) | 1 | 0
Hernia pain (General disorders) | 1 | 0
Hyperthermia (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Infusion site reaction (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Discomfort (General disorders) | 0 | 1
Local swelling (General disorders) | 0 | 1
Secretion discharge (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 12 | 6
Upper respiratory tract infection (Infections and infestations) | 8 | 0
Respiratory tract infection (Infections and infestations) | 6 | 3
Urinary tract infection (Infections and infestations) | 4 | 0
Lower respiratory tract infection (Infections and infestations) | 3 | 1
Oral candidiasis (Infections and infestations) | 3 | 3
Sepsis (Infections and infestations) | 2 | 2
Bronchitis (Infections and infestations) | 2 | 1
Candida infection (Infections and infestations) | 2 | 1
Conjunctivitis (Infections and infestations) | 2 | 0
Herpes zoster (Infections and infestations) | 2 | 0
Paronychia (Infections and infestations) | 2 | 1
Oral herpes (Infections and infestations) | 2 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 1
Fungal infection (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 1
Rhinitis (Infections and infestations) | 1 | 1
Appendicitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Listeriosis (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 1 | 0
Mucosal infection (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 1 | 0
Vaginal infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1
Lymphangitis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Incision site erythema (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Neutrophil count decreased (Investigations) | 14 | 3
White blood cell count decreased (Investigations) | 8 | 1
Weight decreased (Investigations) | 7 | 4
Blood creatinine increased (Investigations) | 3 | 1
Alanine aminotransferase increased (Investigations) | 3 | 1
Electrocardiogram QT prolonged (Investigations) | 3 | 0
Haemoglobin decreased (Investigations) | 2 | 1
Activated partial thromboplastin time prolonged (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 0
Blood magnesium decreased (Investigations) | 2 | 0
Lymphocyte count decreased (Investigations) | 2 | 0
Platelet count decreased (Investigations) | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Blood albumin decreased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Blood iron decreased (Investigations) | 1 | 0
Blood phosphorus decreased (Investigations) | 1 | 0
Blood sodium decreased (Investigations) | 1 | 0
Breath sounds abnormal (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Urine analysis abnormal (Investigations) | 1 | 0
Weight increased (Investigations) | 1 | 0
Blood creatine increased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 34 | 8
Dehydration (Metabolism and nutrition disorders) | 9 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypovitaminosis (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Starvation (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 12 | 1
Dysgeusia (Nervous system disorders) | 9 | 3
Headache (Nervous system disorders) | 7 | 2
Paraesthesia (Nervous system disorders) | 6 | 1
Neuropathy peripheral (Nervous system disorders) | 4 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 0
Syncope (Nervous system disorders) | 2 | 1
Hemiparesis (Nervous system disorders) | 2 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 0
Memory impairment (Nervous system disorders) | 2 | 0
Polyneuropathy (Nervous system disorders) | 2 | 0
Neurotoxicity (Nervous system disorders) | 1 | 1
Presyncope (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 1 | 1
Amnesia (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Paresis (Nervous system disorders) | 1 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Sinus headache (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0
Motor dysfunction (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 5 | 0
Insomnia (Psychiatric disorders) | 5 | 5
Anxiety (Psychiatric disorders) | 2 | 2
Delirium (Psychiatric disorders) | 2 | 0
Agitation (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Irritability (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0
Anorexia nervosa (Psychiatric disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Incontinence (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Renal venous congestion (Renal and urinary disorders) | 1 | 0
Urinary hesitation (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Hypertonic bladder (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Bartholin's cyst (Reproductive system and breast disorders) | 1 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1
Breast tenderness (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 23 | 13
Rash (Skin and subcutaneous tissue disorders) | 10 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 3
Nail discolouration (Skin and subcutaneous tissue disorders) | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 3 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 1 | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 0
Nail toxicity (Skin and subcutaneous tissue disorders) | 2 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 2 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Plantar erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 2 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatosis (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Onychalgia (Skin and subcutaneous tissue disorders) | 0 | 1
Pain management (Surgical and medical procedures) | 1 | 0
Hypotension (Vascular disorders) | 7 | 2
Orthostatic hypotension (Vascular disorders) | 3 | 0
Hypertension (Vascular disorders) | 2 | 1
Phlebitis (Vascular disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 2
Embolism (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 1 | 0
Ischaemia (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-03-02): https://cdn.clinicaltrials.gov/large-docs/16/NCT02387216/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/16/NCT02387216/SAP_001.pdf